CLINICAL TRIAL: NCT00854321
Title: One Centre Follow-up Study on Safety and Efficacy
Brief Title: Patients With Rheumatoid Arthritis (RA) Treated With Rituximab in Kuopio University Hospital
Acronym: KuoRituxi1
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Oili Kaipiainen-Seppänen, Kuopio University Hospital
Other Study IDs: KuoRituxi1
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-03

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; rituximab; therapy
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with active RA: drug, follow-up
  Interventions: Drug: rituximab; Drug: rituximab, observational study amon patients with active RA

INTERVENTIONS:
Drug: rituximab — rituximab two 1000 mg intravenous infusions separated by two weeks
Drug: rituximab, observational study amon patients with active RA — two 1000 mg intravenous infusions separated by 2 weeks

SUMMARY:
One centre follow-up study on safety and efficacy of treatment with rituximab among patients with RA during 4 year period. Basic data is collected for the national register of biologicals.

DETAILED DESCRIPTION:
Data is collected on regular visits in the outpatient department. In collection national register forms have been used.

ELIGIBILITY:
Inclusion Criteria:

* active RA without response to earlier treatment

Exclusion Criteria:

* contraindications to rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with active RA in one centre
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2004-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
ACR20 ACR50 ACR70 response | 6 and 12 months

SECONDARY OUTCOMES:
Duration of clinical response | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Oili Kaipiainen-Seppänen, MD, Study Director — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

REFERENCES:
- [Background] Keystone E, Burmester GR, Furie R, Loveless JE, Emery P, Kremer J, Tak PP, Broder MS, Yu E, Cravets M, Magrini F, Jost F. Improvement in patient-reported outcomes in a rituximab trial in patients with severe rheumatoid arthritis refractory to anti-tumor necrosis factor therapy. Arthritis Rheum. 2008 Jun 15;59(6):785-93. doi: 10.1002/art.23715. PMID 18512710